CLINICAL TRIAL: NCT02871596
Title: Effect of a Proprietary Dietary Supplement on Fecal Volatile Organic Compounds - a Randomized, Placebo-controlled, Double-blind, Cross-over Study
Brief Title: Effect of a Proprietary Dietary Supplement on Fecal Volatile Organic Compounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Utah State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 16-PHX-0003
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Healthy
MeSH Terms: interventions — Flavonoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo,Flavonoids,Flavonoids+Prebiotics (Experimental): Participants will receive three treatments, for three weeks each, with 21 day washout period between each product.
  Interventions: Other: Placebo; Dietary Supplement: Flavonoids; Dietary Supplement: Flavonoids+Prebiotics
- Placebo,Flavonoids+Prebiotics,Flavonoids (Experimental): Participants will receive three treatments, for three weeks each, with 21 day washout period between each product.
  Interventions: Other: Placebo; Dietary Supplement: Flavonoids; Dietary Supplement: Flavonoids+Prebiotics
- Flavonoids,Placebo,Flavonoids+Prebiotics (Experimental): Participants will receive three treatments, for three weeks each, with 21 day washout period between each product.
  Interventions: Other: Placebo; Dietary Supplement: Flavonoids; Dietary Supplement: Flavonoids+Prebiotics
- Flavonoids,Flavonoids+Prebiotics,Placebo (Experimental): Participants will receive three treatments, for three weeks each, with 21 day washout period between each product.
  Interventions: Other: Placebo; Dietary Supplement: Flavonoids; Dietary Supplement: Flavonoids+Prebiotics
- Flavonoids+Prebiotics,Placebo,Flavonoids (Experimental): Participants will receive three treatments, for three weeks each, with 21 day washout period between each product.
  Interventions: Other: Placebo; Dietary Supplement: Flavonoids; Dietary Supplement: Flavonoids+Prebiotics
- Flavonoids+Prebiotics,Flavonoids,Placebo (Experimental): Participants will receive three treatments, for three weeks each, with 21 day washout period between each product.
  Interventions: Other: Placebo; Dietary Supplement: Flavonoids; Dietary Supplement: Flavonoids+Prebiotics

INTERVENTIONS:
Other: Placebo — A combination of maltodextrins and red and blue food colors.
Dietary Supplement: Flavonoids — A combination of blueberry extract, black current extract, and black rice extract.
Dietary Supplement: Flavonoids+Prebiotics — A combination of blueberry extract, black current extract, black rice extract, inulin, and fructooligosaccharide.

SUMMARY:
The purpose of the study is to determine the effects of both an anthocyanin-rich polyphenol blend and an anthocyanin-rich polyphenol blend combined with a prebiotic blend on fecal microbiota metabolism (assessed by gas chromatograph - mass spectrometry (GC-MS) headspace analysis) and fecal microbiota composition (assessed by next generation sequencing).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race or ethnicity between 18 to 70 years of age, inclusive;
* Body mass index (BMI) between 20 - 32 inclusive;
* Non-smoking status;
* Willing to consume assigned dietary supplements for a total of 6 weeks;
* Have access to email and a digital camera or camera phone.

Exclusion Criteria:

* Age <18 or >70 years;
* BMI <20 or >32;
* Uncontrolled hypertension defined as diastolic blood pressure ≥95 mm Hg or systolic blood pressure ≥160 mm Hg;
* Self-reported presence of atherosclerotic disease and/or cardiopulmonary disease;
* Renal, hepatic, endocrine, gastrointestinal or other systemic disease;
* For women, pregnancy, breast feeding or postpartum less than 6 months;
* Current participation in another research study;
* Allergy to the components in the dietary supplement (inulin, fructooligosaccharide, blueberries, black currant, rice);
* History of drug or alcohol abuse;
* Use of antibiotics within the last 6 months;
* Use of prebiotics or flavonoid-containing dietary supplements within the last 30 days;
* Multiple food allergies or significant food preferences or restrictions that would interfere with diet adherence;
* Chronic use of over-the-counter medication which would interfere with study endpoints including NSAIDS, laxatives and antacids;
* Participating in or planning to begin a weight loss diet during the study period;
* Lifestyle or schedule incompatible with the study protocol;
* Other medical, psychiatric, or behavioral conditions that in the view of the principal investigator may present a safety hazard to the participant or interfere with study participation or the ability to follow the intervention protocol;
* Use of tobacco products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fecal volatile methyl sulfides at day 21, day 63, day 105 | baseline, day 21, day 63, day 105
  assessed by gas chromatograph - mass spectrometry (GC-MS) headspace analysis

SECONDARY OUTCOMES:
Change from baseline in all fecal VOCs at day 21, day 63, day 105 | baseline, day 21, day 63, day 105
Change from baseline fecal short chain fatty acids at day 21, day 63, day 105 | baseline, day 21, day 63, day 105
Change from baseline fecal microbiota composition at day 21, day 63, day 105 | baseline, day 21, day 63, day 105

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lefevre, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No